CLINICAL TRIAL: NCT07021950
Title: Ivonescimab (AK112) Plus FOLFIRI Versus Bevacizumab Plus FOLFIRI as Second-line Treatment of MSS/pMMR Metastatic Colorectal Cancer: a Randomized, Controlled, Multicenter Phase II Study
Brief Title: AK112 Plus FOLFIRI Versus Bevacizumab Plus FOLFIRI as Second-line Treatment of MSS/pMMR Metastatic Colorectal Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Rui-hua Xu, MD, PhD, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AK112-CRC
Record Dates: First submitted 2025-06-06; First posted 2025-06-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Colorectal Cancer; Ivonescimab
MeSH Terms: conditions — Colorectal Neoplasms | interventions — IFL protocol; Bevacizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AK112+FOLFIRI (Experimental): experimental group receives AK112 at 20 mg/kg via intravenous infusion on day 1 of each cycle (Q2W) combined with FOLFIRI chemotherapy (Q2W)
  Interventions: Drug: AK112; Drug: FOLFIRI
- bevacizumab+FOLFIRI (Active Comparator): Control group receives bevacizumab at 5 mg/kg via intravenous infusion on day 1 of each cycle (Q2W) combined with FOLFIRI chemotherapy (Q2W)
  Interventions: Drug: FOLFIRI; Drug: Bevacizumab

INTERVENTIONS:
Drug: AK112 — AK112：20mg/kg，Q2W。Administered over 60 minutes (±10 minutes). For intolerable cases, infusion duration may extend up to 120 minutes. During treatment, dosing delays are allowed for up to 12 weeks (calculated from the last dose). AK112 may be resumed after 12 weeks under the following conditions: If treatment is paused due to glucocorticoid tapering for managing immune-related adverse events (irAEs);If treatment is paused due to adverse events unrelated or deemed unrelated to AK112; Resumption is permitted only if the investigator judges continued therapy beneficial, following discussion with relevant medical personnel.
  Other Names: Ivonescimab
  Arms: AK112+FOLFIRI
Drug: FOLFIRI — FOLFIRI：Irinotecan, 180 mg/m² IV over 30-90 minutes (Day 1); Leucovorin (LV), 400 mg/m² IV over 2 hours (Day 1); 5-FU, 400mg/m²IV Day1, then 1200 mg/(m².d) ×2 days (total 2400 mg/m² ,IV over 46-48 hours).Q2W.
Drug: Bevacizumab — Bevacizumab：5 mg/kg，Q2W. The initial intravenous infusion should last approximately 90 minutes. If the first infusion is well tolerated, the duration of the second infusion can be reduced to approximately 60 minutes. Should the participant also tolerate the 60-minute infusion well, then all subsequent infusions may be administered over a period of approximately 30 minutes. Continuous monitoring for potential infusion-related reactions during the drip is required; if an infusion-related reaction occurs, the infusion rate should be promptly reduced or the infusion temporarily halted.
  Arms: bevacizumab+FOLFIRI

SUMMARY:
This study is a multicenter, open-label phase II trial conducted to assess the safety and antitumor activity of Ivonescimab (AK112) plus FOLFIRI versus bevacizumab plus FOLFIRI as second-line treatment in subjects with MSS/pMMR metastatic colorectal cancer who have experienced intolerance to oxaliplatin-containing first-line therapy or disease progression, or recurrence within 6 months after oxaliplatin adjuvant therapy.

DETAILED DESCRIPTION:
After obtaining informed consent, the experimental group receives AK112 at 20 mg/kg via intravenous infusion on day 1 of each cycle (Q2W) combined with FOLFIRI chemotherapy (Q2W), while the control group receives bevacizumab at 5 mg/kg via intravenous infusion on day 1 of each cycle (Q2W) in combination with FOLFIRI (Q2W). Treatment continues until disease progression, death, intolerable toxicity, withdrawal of consent, initiation of new antitumor therapy, or other protocol-specified reasons for discontinuation. The maximum treatment duration is 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign written informed consent
2. Agree to provide tumor and blood samples for biomarker detection
3. Age ≥18 and ≤75 years at enrollment, regardless of gender
4. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1
5. Expected survival ≥3 months
6. Pathologically confirmed locally advanced unresectable or metastatic colorectal adenocarcinoma
7. Confirmed MSS/pMMR-type CRC by immunohistochemistry (IHC), PCR, or NGS
8. Intolerance to oxaliplatin-containing standard first-line therapy, disease progression, or recurrence within < 6 months after oxaliplatin adjuvant therapy
9. Adequate organ function (last 14 days without intervention):

   1. Absolute neutrophil count (ANC) ≥1.5×10⁹/L without granulocyte colony-stimulating factor1.
   2. Platelets ≥100×10⁹/L without transfusion1.
   3. Hemoglobin >9 g/dL without transfusion or erythropoietin1.
   4. Total bilirubin ≤1.5×ULN1.
   5. AST/ALT ≤2.5×ULN1.
   6. Serum creatinine ≤1.5×ULN and creatinine clearance (Cockcroft-Gault) ≥60 mL/min1.
   7. INR or PT ≤1.5×ULN1.
   8. Normal thyroid function (TSH within normal range; if TSH abnormal, FT3/FT4 must be normal)1.
10. For HBV/HCV-infected subjects:Chronic HBV: Undetectable viral load under suppressive therapy if required; HCV: Stable status; ongoing antiviral therapy must continue if applicable;Co-infection of HBV and HCV is excluded (prior HCV infection with negative RNA is acceptable)
11. Females of childbearing potential: Negative pregnancy test (urine/serum) within 3 days prior to first dose. Effective contraception from screening until 120 days after last dose
12. Non-sterilized males: Effective contraception from screening until 120 days after last dose Willing and able to comply with study visits, treatment, and procedures

Exclusion Criteria:

* 1.Known as MSI-H or dMMR status 2.History of or concurrent malignancies within 3 years, except cured local tumors (e.g., basal cell skin cancer, squamous cell skin cancer, superficial bladder cancer, cervical carcinoma in situ) 3.Current or prior central nervous system (CNS) or leptomeningeal metastases 4.Proteinuria ≥2+ on dipstick/urinalysis or 24-hour urine protein ≥1.0 g (patients with 1+ proteinuria require confirmation via 24-hour urine collection) 5.Unresolved toxicities from prior therapy exceeding NCI CTCAE v5.0 Grade 1 (except alopecia or neuropathy ≤Grade 2) 6.Gastrointestinal perforation ≤1 year before enrollment or a history of GI perforation 7.Prior irinotecan treatment (including irinotecan injection or liposomal irinotecan) 8.Prior anti-angiogenic small molecule targeted therapy (e.g., fruquintinib) 9.Concurrent participation in an interventional clinical trial or use of investigational drugs/devices ≤4 weeks before the first dose 10.Current or prior non-infectious pneumonitis or interstitial lung disease requiring systemic corticosteroids 11.Active autoimmune disease requiring systemic therapy within 2 years (e.g., disease-modifying agents, corticosteroids, immunosuppressants). Replacement therapy (e.g., thyroxine, insulin) is permitted 12.History of immunodeficiency, positive HIV antibody test, or long-term use of systemic corticosteroids/immunosuppressants (short-term steroids for COPD or allergies allowed) 13.Active tuberculosis (confirmed or suspected requiring exclusion) or syphilis infection 14.Severe infection (e.g., sepsis, pneumonia requiring hospitalization) ≤4 weeks before the first dose or active infection requiring systemic anti-infectives ≤2 weeks (excluding HBV/HCV antivirals) 15.Significant bleeding history (e.g., hemoptysis ≥1 teaspoon of blood, gastrointestinal bleeding) ≤1 month or antiplatelet/anticoagulant therapy ≤10 days before the first dose 16.Active/past inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis, chronic diarrhea) 17.Uncontrolled comorbidities (e.g., metabolic disorders, peptic ulcers, psychiatric conditions affecting compliance) 18.Cardiac history: myocardial infarction, NYHA Class ≥2 heart failure, unstable angina ≤12 months; arterial/venous thromboembolism ≤6 months; uncontrolled hypertension (SBP >150 mmHg or DBP >90 mmHg) 19.Prior immune therapy (checkpoint inhibitors, CAR-T, etc.) targeting tumor immunity 20.Major surgery ≤30 days before/after the first dose or minor surgery ≤3 days before the first dose (excluding IV catheter placement) 21.Live/attenuated vaccines ≤30 days before the first dose or planned during the study; inactivated vaccines permitted 22.History of allogeneic organ or hematopoietic stem cell transplantation 23.Hypersensitivity to study drug components or monoclonal antibodies 24.History of psychiatric disorders, substance abuse, or alcoholism 25.Pregnancy or lactation 26.Any current or past disease, therapy, or abnormal laboratory finding that may confound study results, interfere with full study participation, or compromise the participant's best interest by continuing in the study Conditions that may confound results or pose undue risk (e.g., leukemoid reaction (WBC >20×10⁹/L), ≥10% weight loss ≤3 months)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2025-08-10 (Estimated); Primary Completion 2027-10-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
PFS | up to 24 months
  Refers to the date from the date of admission to the date of the first progression of disease or death of any cause, using Response Evaluation Criteria in Solid Tumors version 1.1(RECIST v1.1)

SECONDARY OUTCOMES:
ORR | up to 24 months
  The proportion of patients achieving complete response (CR) or partial response (PR) as their best overall response per RECIST v1.1 criteria.
DCR | up to 24 months
  The proportion of patients achieving CR, PR, or stable disease (SD) lasting for ≥ a prespecified duration
DoR | up to 24 months
  monitor the length of time patients experience a reduction in tumor size orstabilization of disease following the treatment
OS | up to 3 years
  The time interval between the start date of study drug and the date of death (any cause)
AE | up to 36 months untill study complete
  Number and percentage of participants with adverse events(AEs)

CONTACTS AND LOCATIONS:
Overall Officials: Ruihua Xu, MD, PhD, Principal Investigator — Sun Yat-sen University